CLINICAL TRIAL: NCT02759250
Title: A Pilot, Phase Ib Feasibility Study of ARGX-110 in Patients With Nasopharyngeal Carcinoma (NPC)
Brief Title: A Study of ARGX-110 in Patients With Nasopharyngeal Carcinoma (NPC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARGX-110-1401
Record Dates: First submitted 2016-04-22; First posted 2016-05-03 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- adjuvant monotherapy (Experimental): ARGX-110 5mg/kg once every three weeks for a maximum of 18 cycles
  Interventions: Drug: ARGX-110
- metastatic/recurrent monotherapy (Experimental): ARGX-110 5mg/kg once every three weeks until disease progression
  Interventions: Drug: ARGX-110
- metastatic/recurrent combination therapy (Experimental): ARGX-110 5mg/kg once every three weeks plus chemotherapy until disease progression. The choice of the chemotherapy agents is limited to: cisplatin, carboplatin, 5-fluorouracil, gemcitabine and paclitaxel.
  Interventions: Drug: ARGX-110

INTERVENTIONS:
Drug: ARGX-110

SUMMARY:
To characterize the safety profile of ARGX-110 administered as mono- or combination therapy to patients with NPC at various stages of its natural history (adjuvant vs. metastatic).

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years.
* Written informed consent prior to any study-related procedure
* Willing and able to comply with protocol-specified procedures and scheduled evaluations
* Pathological diagnosis of nasopharyngeal carcinoma (NPC)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1or 2
* Absolute neutrophil count (ANC) > 0.5 x 109/L
* Haemoglobin > 80 g/L
* Platelet count ≥ 50 x 109/L
* Total bilirubin ≤ 2 x the upper limit of normal (ULN)
* Alanine transaminase (ALT) ≤ 5 x ULN
* Serum creatinine ≤ 2 x ULN

Exclusion criteria:

* History or clinical evidence of neoplastic central nervous system (CNS) involvement. Note: Irradiated brain metastases that have been stable for > 1 month and do not require systemic glucocorticoid administration are allowed
* Major surgery within 4 weeks of ARGX-110 first dose administration
* Unresolved grade 3 or 4 toxicity from prior therapy (except mucositis from local radiation therapy).
* Active, untreated viral, bacterial, or systemic fungal infection
* Childbearing potential unless using an adequate measure of contraception
* Pregnancy or lactation. History of hypersensitivity to recombinant proteins
* Any clinical finding, including psychiatric and behavioural problems, which, in the opinion of the Investigator, precludes the patient from safely participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-02; Primary Completion 2018-04-25 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Incidence and grading of AEs | measured at screening, Day 1, Day 8, Day 15, Day 42, thereafter every 42 days until Day 378
  Change from baseline in incidence and grading of AEs according to the Common Terminology Criteria for Adverse Event (NCI-CTCAE) Version 4.03

SECONDARY OUTCOMES:
Pharmacokinetic profile of ARGX110 by Cmax | measured at Day 1 pre and post dose, Day 8, Day 15, Day 42 pre and post dose and thereafter every 42 days until Day 378
  Change from baseline in Measurement of drug concentration in the blood
Pharmacokinetic profile of ARGX110 by AUC | measured at Day 1 pre and post dose, Day 8, Day 15, Day 42 pre and post dose and thereafter every 42 days until Day 378
  Change in Measurement of drug concentration in the blood
Biomarkers CD70 immunohistochemistry (IHC) | measured at Screening, Day 42, and thereafter every 42 days until day Day 378
  Change in Measurement of concentration in tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Rottey, MD, Principal Investigator — UZG - Universitair Ziekenhuis Gent
Locations (1):
- UZG - Universitair Ziekenhuis Gent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided